CLINICAL TRIAL: NCT04506047
Title: Acute and Long-term Outcomes of Patients Presenting With Acute Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention
Brief Title: Acute and Long-term Outcomes of Patients With Acute Myocardial Infarction Treated With PCI
Acronym: SINERGY-ACUTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Institute of Cardiovascular Diseases, Vojvodina (Other); Clinical Hopital Center Zemun (Unknown); University Hospital Medical Center Bezanijska Kosa (Unknown); Clinical Centre of Kragujevac (Unknown); Clinical Hospital Center Zvezdara (Unknown)
Responsible Party: Principal Investigator, Goran Stankovic, Professor, Clinical Centre of Serbia
Other Study IDs: 570/11
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Acute Myocardial Infarction; Coronary Artery Disease
Keywords: AMI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Myocardial Infarction: Consecutive patients with acute myocardial infarction
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Percutaneous Coronary Intervention

SUMMARY:
Randomized studies may often be burdened by the selective nature of patient inclusion thus not reflecting real-world outcomes. This is evident from the discrepancy in the mortality rates reported in major randomized trials enrolling patients with acute myocardial infarction (AMI), as compared with registry data.

The primary objective of this observational study is to assess short- and long-term outcomes of unselected, real-world patients presenting with AMI and treated with contemporary percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction referred to catheterization laboratory for percutaneous coronary intervention

Exclusion Criteria:

* Initial acute myocardial infarction diagnosis not confirmed
* Patients with acute myocardial infarction not undergoing invasive coronary angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry is based on consecutive patients with the initial diagnosis of acute myocardial infarction on admission to hospital, who are referred to invasive treatment, i.e. invasive coronary angiography with an intention to perform percutaneous coronary intervention. The study population will include both retrospective, multi-center registry data starting with the year 2009, and the prospectively enrolled patients according to the same pre-specified, broad inclusion/exclusion criteria. The underlying intention is to short- and long-term outcomes of a large population of unselected, real-world patients presenting with AMI and treated with PCI.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 1 year
  Rate of all-cause mortality at 1 year

SECONDARY OUTCOMES:
Rate of all-cause mortality | 5 years
  Rate of all-cause mortality at 5 years
Rate of cardiovascular mortality | 5 years
  Rate of cardiovascular mortality at 5 years

OTHER OUTCOMES:
Rate of myocardial infarction | 5 years
  Rate of myocardial infarction at 5 years
Rate of repeat revascularization | 5 years
  Rate of repeat revascularization at 5 years
Rate of stroke | 5 years
  Rate of stroke at 5 years
Rate of new or worsening heart failure | 5 years
  Rate of new or worsening heart failure at 5 years
Rate of new or worsening heart failure | 1 year
  Rate of new or worsening heart failure at 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Centre of Serbia, Department of Cardiology, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided